CLINICAL TRIAL: NCT06404892
Title: ARISCAT, ASA and LAS VEGAS Risk Scores and the Incidence of Postoperative Pulmonary Complications in Patients Undergoing Thoracic Surgery With Single-lung Ventilation
Brief Title: ARISCAT, ASA and LAS VEGAS Risk Scores and the Incidence of Postoperative Pulmonary Complications in Thoracic Surgery
Status: Recruiting | Type: Observational
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Principal Investigator, Andre Prato Schmidt, Anesthesiologist, Hospital Nossa Senhora da Conceicao
Other Study IDs: 75871723.4.0000.5530
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Complications
Keywords: postoperative pumonary complications; ARISCAT score; LAS VEGAS score; ASA score
MeSH Terms: conditions — Postoperative Complications | interventions — One-Lung Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients undergoing thoracic surgery and single-lung ventilation.
  Interventions: Procedure: Single-lung ventilation

INTERVENTIONS:
Procedure: Single-lung ventilation — Patients undergoing thoracic surgery and intraoperative single-lung ventilation.

SUMMARY:
Postoperative pulmonary complications (PPC) are among the main complications after the anesthetic-surgical procedure. It can be said that thoracic surgery results in impaired respiratory function in the postoperatively, due to the decrease in lung volumes and capacities (the vital capacity decreases by approximately 50-60% and functional residual capacity decreases by approximately 30% in the first 24 hours after surgery) diaphragm dysfunction, gas exchange impaired, cough and ineffective mucociliary clearance. Thus, our hypothesis is that the application of preoperative risk scores normally used for non-cardiac and non-thoracic surgeries may be effective on the predictability of the occurrence of CPP in patients undergoing ventilation single-lung. This is a prospective observational study in order to evaluate the performance of the ASA, ARISCAT and LAS VEGAS risk scores for predict the occurrence of postoperative pulmonary complications (PPC) in patients undergoing thoracic surgery with single-lung ventilation.

DETAILED DESCRIPTION:
Postoperative pulmonary complications (PPC) are among the main complications after the anesthetic-surgical procedure; CPP prolong hospital stay and increase costs in health systems. It can be said that thoracic surgery results in impaired respiratory function in the postoperatively, due to the decrease in lung volumes and capacities (the vital capacity decreases by approximately 50-60% and functional residual capacity decreases by approximately 30% in the first 24 hours after surgery) diaphragm dysfunction, gas exchange impaired, cough and ineffective mucociliary clearance.

Thus, our hypothesis is that the application of preoperative risk scores normally used for non-cardiac and non-thoracic surgeries may be effective in the predictability of the occurrence of CPP in patients undergoing ventilation single-lung. In this study, we will prospectively evaluate the performance of ASA, ARISCAT and LAS VEGAS scores in predicting patients who present with CPP in thoracic surgeries using single-lung ventilation. We will also analyze other potential patient risk factors as well as complications presented.

This is a prospective observational study. Data will be collected using a standardized form at the surgical center of Hospital Nossa Senhora da Conceição and at the Hospital de Clínicas de Porto Alegre, evaluated preoperatively, intraoperatively and postoperatively. Direct observation and recording of variables studied by the anesthesiology medical team of both hospitals, previously trained and supervised by the main researcher. Patients will be monitored until hospital discharge or up to a maximum period of 30 days of hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing any thoracic procedure associated with intraoperative single-lung ventilation.

Exclusion Criteria:

* Patients undergoing cardiac surgery, pregnant women, patient refusal, contraindications to proposed surgical, anesthetic or analgesic techniques, sepsis, psychiatric illness, uncontrolled endocrine, kidney or liver disease and coagulopathies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing any thoracic procedure associated with intraoperative use of single-lung ventilation.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | up to 30 days after surgery
  Incidence of composite pulmonary complications after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Andre P Schmidt, MD, Principal Investigator — Hospital Nossa Senhora da Conceição
Locations (1):
- HCPA, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No